CLINICAL TRIAL: NCT05903027
Title: Effectiveness and Tolerability of Rimegepant as Acute Migraine Treatment: a Prospective, Multicentric, Cohort Study (GAINER)
Brief Title: Gepant treAtments: EffectIveNess and tolERability (GAINER)
Acronym: GAINER
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Società Italiana per lo Studio delle Cefalee (Other); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Università degli Studi dell'Aquila (Other); University of Roma La Sapienza (Other); Azienda Ospedaliero Universitaria Policlinico Modena (Other); Ospedale di Piove di Sacco (Unknown); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); A.O.U. Città della Salute e della Scienza (Other); Cliniche Humanitas Gavazzeni (Other); University of Campania Luigi Vanvitelli (Other); Ospedale Santo Stefano (Other); Azienda Policlinico Umberto I (Other); Auxologico San Luca (Other); Asst Degli Spedali Civili Di Brescia (Other); Carlo Besta Neurological Institute (Other)
Responsible Party: Principal Investigator, Luigi Francesco Iannone, Researcher, University of Florence
Other Study IDs: RICe_1
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura; Chronic Migraine
Keywords: Headache; Medication overuse headache; Pain; Gepant; Triptan
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache; Headache Disorders, Secondary; Pain | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic migraine: Patients affected by an episodic pattern migraine(< 15 monthly headache days) with or without aura according to ICHD-III criteria.
  Interventions: Drug: Rimegepant 75 MG Disintegrating Oral Tablet
- Chronic migraine: Patients affected by chronic migraine according to ICHD-III criteria.
  Interventions: Drug: Rimegepant 75 MG Disintegrating Oral Tablet

INTERVENTIONS:
Drug: Rimegepant 75 MG Disintegrating Oral Tablet — Patients using Rimegepant 75 mg orally disintegrating tablet to treat acute migraine attacks

SUMMARY:
The purpose of this prospective and multicentric study is to evaluate the effectiveness and tolerability of rimegepant as acute migraine treatment in a cohort of episodic or chronic migraine patients.

DETAILED DESCRIPTION:
Rimegepant belongs to the gepants family, small molecules calcitonin gene-related peptide (CGRP) receptor antagonists. It is a new generation gepants, currently available as an orally disintegrating tablet at a single dose of 75 mg. It has a double indication both for acute treatment for migraine with and without aura and preventive treatment of episodic migraine. Previous randomized, placebo-controlled phase 3 trials and open label extensions demonstrated its effectiveness in the acute setting for a single migraine attack of both the oral tablet and the orally disintegrating tablet. Pooled analysis of previous randomized clinical trials also showed rimegepant effectiveness in patients with a history of insufficient response to triptans.

Previous studies also demonstrated a good tolerability profile. The most commonly reported adverse events were nausea, nasopharyngitis, upper respiratory tract infections and urinary tract infection.

In this prospective multicentric study we aim to evaluate Rimegepant effectiveness and tolerability as acute migraine treatment in a real-world setting.

Subjects who meet the inclusion criteria will be enrolled and will participate in the study. Baseline demographic and clinical data will be collected at the baseline. Patients will be asked to treat their next migraine attack with Rimegepant 75 mg orally disintegrating tablet.

Data will be collected at baseline, during at least 4 migraine attacks treated with Rimegepant and at 3 months follow-up.

Subjects will be asked to complete assessment of their migraine attack at baseline and at 30 - 60 - 90 and 120 minutes after administration of the acute treatment for at least four migraine attacks. A final timepoint at 24 hours post-dose will be assessed only for the first attack.

Data collection will focus on: i) demographic data, ii) migraine history, iii) pain level and evolution, iv) presence and evolution of migraine associated symptoms, most bothersome symptom and aura, v) migraine associated disability, vi) patients's global impression of change (PGIC) and evaluation on the acute treatment (Migraine-ACT), vii) tolerability and eventual treatment-emergent adverse events. The online database REDCap will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the 3rd edition of the International Classification of Headache Disorder (ICHD-III).
* At least 3 MMDs
* Good compliance to study procedures
* Availability of headache diary at least of the preceding months before enrollment

Exclusion Criteria:

* Subjects with contraindications for use of gepants;
* Concomitant diagnosis of medical diseases and/or comorbidities that, in the Investigator's opinion might interfere with study assessments;
* medical comorbidities that could interfere with study results;
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric study on patients attending the outpatient clinic of Italian Headache centres who meet criteria for Rimegepant use for acute migraine treatments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Headache pain freedom at 2 hours post-dose during the first attack | 2 hours post-dose
  The percentage of subjects that report no headache pain at 2 hours after drug intake. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Occurrence of treatment-emergent adverse events | 12 weeks
  To evaluate the safety and tolerability of Rimegepant in migraine subjects.

SECONDARY OUTCOMES:
Headache pain freedom at 2 hours post-dose across all treated attacks | 2 hours post-dose for all treated attacks
  The percentage of subjects that report no headache pain at 2 hours after drug intake across all' treated attacks. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Headache pain relief at 2 hours post-dose during the first attack | 2 hours post-dose
  The percentage of subjects that report mild or none headache pain at 2 hours after drug intake during the first attack. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Headache pain relief at 2 hours post-dose across all treated attacks | 2 hours post-dose for all treated attacks
  The percentage of subjects that report mild or none headache pain at 2 hours after drug intake across all treated attack. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Ability to function normally at 2 hours post-dose during the first attack | 2 hours post-dose
  The percentage of subjects that self-report no functional disability at 2 hours post-dose. Functional disability will be assessed through the Functional Disability Scale (FDS), a four-point scale: normal, mildly impaired, severely impaired, requires daily activities interruption.
Ability to function normally at 2 hours post-dose across all treated attacks | 2 hours post-dose for all treated attacks
  The percentage of subjects that self-report no functional disability at 2 hours post-dose. Functional disability will be assessed through the Functional Disability Scale, a four-point scale: normal, mildly impaired, severely impaired, requires daily activities interruption.
Freedom from the most bothersome symptom (MBS) associated with migraine at 2 hours post-dose during the first attack | 2 hours post-dose
  The percentage of subjects that report complete MBS resolution at 2 hours after drug intake. MBS will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Headache recurrence for the first-attack | between 2 hours and 24 hours post-dose
  Percentage of subjects who became pain free at 2 hours post-dose and report new headache pain within 24 hours post-dose.
Rescue medications use for the first attack | between 2 hours and 24 hours post dose
  Percentage of subjects who take a rescue medication after 2 hour post-dose. Rescue medications will be measured using a binary scale (0=no consumption, 1=consumption)
Treatment satisfaction | 2 hours post-dose for all treated attacks
  Level of patients' self-reported satisfaction which will be measured on a 0-10 visual analogue scale (0=no satisfaction, 10= the highest satisfaction) and Patients Global Impression of Change (0= no changing, 7= a change that makes the difference).
Self-reported treatment effectiveness | 12 weeks
  Level of patients' self-reported treatment effectiveness measured by Migraine Assessment of Current Therapy (Migraine-ACT) a 4-item questionnaire about treatment effectiveness and daily life repercussions.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - SOD Centro Cefalee e Farmacologia Clinica, AOU Careggi, Florence
  - IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lipton RB, Croop R, Stock EG, Stock DA, Morris BA, Frost M, Dubowchik GM, Conway CM, Coric V, Goadsby PJ. Rimegepant, an Oral Calcitonin Gene-Related Peptide Receptor Antagonist, for Migraine. N Engl J Med. 2019 Jul 11;381(2):142-149. doi: 10.1056/NEJMoa1811090. PMID 31291516
- [Background] Croop R, Goadsby PJ, Stock DA, Conway CM, Forshaw M, Stock EG, Coric V, Lipton RB. Efficacy, safety, and tolerability of rimegepant orally disintegrating tablet for the acute treatment of migraine: a randomised, phase 3, double-blind, placebo-controlled trial. Lancet. 2019 Aug 31;394(10200):737-745. doi: 10.1016/S0140-6736(19)31606-X. Epub 2019 Jul 13. PMID 31311674
- [Background] Lipton RB, Blumenfeld A, Jensen CM, Croop R, Thiry A, L'Italien G, Morris BA, Coric V, Goadsby PJ. Efficacy of rimegepant for the acute treatment of migraine based on triptan treatment experience: Pooled results from three phase 3 randomized clinical trials. Cephalalgia. 2023 Feb;43(2):3331024221141686. doi: 10.1177/03331024221141686. PMID 36739511
- [Derived] Iannone LF, Vaghi G, Sebastianelli G, Casillo F, Russo A, Silvestro M, Pistoia F, Volta GD, Cortinovis M, Chiarugi A, Montisano DA, Prudenzano MP, Cevoli S, Mampreso E, Avino G, Romozzi M, Valente M, Fasano C, Battistini S, Granato A, Piella EM, Rainero I, Ornello R, De Icco R; Italian Headache Registry (RICe) Study Group. Effectiveness and tolerability of rimegepant in the acute treatment of migraine: a real-world, prospective, multicentric study (GAINER study). J Headache Pain. 2025 Jan 6;26(1):4. doi: 10.1186/s10194-024-01935-8. PMID 39762740